CLINICAL TRIAL: NCT02136082
Title: Asha Improving Health and Nutrition of Indian Women With AIDS and Their Children
Acronym: Asha2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: All India Institute of Medical Sciences (Other); University of California, San Francisco (Other); University of California, Irvine (Other)
Responsible Party: Principal Investigator, Adeline Nyamathi, PhD, Distinguished Professor, University of California, Irvine
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: NIHMS098729
Record Dates: First submitted 2014-05-08; First posted 2014-05-12 (Estimated); Last update posted 2018-10-09 (Actual); Status verified 2018-10

CONDITIONS: HIV Infection
Keywords: HIV; Women; Children; Nutrition
MeSH Terms: conditions — HIV Infections | interventions — Food

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Asha Support + Training (Experimental): Asha Support + Training: 1) Group discussions delivered over a six month period that cover four main categories a) Staying Healthy; b) Caregiving; c) Staying Upbeat; and d) Healthy Eating for Self and Family; 2) Referral for Life Skills Classes to teach women about selling fruit and vegetables and dried fish, sewing and embroidery and computer skills; 3) Asha Support. Women are visited by an Asha to discuss the group sessions, any difficulties the women may be experiencing with staying on ART, and ways to help women stay on the regimen.
  Interventions: Behavioral: Asha Support + Training
- Asha Support + Food (Experimental): Asha Support + Food 1) Group discussions delivered over a six month period that cover three main categories a) Staying Healthy; b) Caregiving; and c) Staying Upbeat; 2) Referral for Life Skills Classes to teach women about selling fruit and vegetables and dried fish, sewing and embroidery and computer skills; 3) Asha Support. Women are visited by an Asha to discuss the group sessions, any difficulties the women may be experiencing with staying on ART, and ways to help women stay on the regimen; 4) Food supplementation of high protein food such as urad dal or tur dal.
  Interventions: Behavioral: Asha Support + Food
- Asha Support + Training + Food (Experimental): Asha Support + Training + Food: 1) Group discussions delivered over a six month period that cover four main categories a) Staying Healthy; b) Caregiving; c) Staying Upbeat; and d) Healthy Eating for Self and Family; 2) Referral for Life Skills Classes to teach women about selling fruit and vegetables and dried fish, sewing and embroidery and computer skills; 3) Asha Support. Women are visited by an Asha to discuss the group sessions, any difficulties the women may be experiencing with staying on ART, and ways to help women stay on the regimen; 4) Food supplementation of high protein food such as urad dal or tur dal.
  Interventions: Behavioral: Asha Support + Training + Food
- Asha Support Only (Active Comparator): Asha Support Only 1) Group discussions delivered over a six month period that cover three main categories a) Staying Healthy; b) Caregiving; c) Staying Upbeat; 2) Referral for Life Skills Classes to teach women about selling fruit and vegetables and dried fish, sewing and embroidery and computer skills; 3) Asha Support. Women are visited by an Asha to discuss the group sessions, any difficulties the women may be experiencing with staying on ART, and ways to help women stay on the regimen.
  Interventions: Behavioral: Asha Support Only

INTERVENTIONS:
Behavioral: Asha Support + Training
  Arms: Asha Support + Training
Behavioral: Asha Support + Food
  Arms: Asha Support + Food
Behavioral: Asha Support + Training + Food
  Arms: Asha Support + Training + Food
Behavioral: Asha Support Only
  Arms: Asha Support Only

SUMMARY:
Building upon the successful qualitative Phase I of the study, Phase II commences in month 10. The Project manager and research staff will recruit 600 women living with AIDS (WLA) and their oldest child between the ages of 3 and 8. The WLA will be recruited from Primary Health Centers (PHCs) randomly selected from 72 closest PHCs in terms of HIV prevalence in the rural Andhra Pradesh (AP) area of Nellore. WLA will be recruited by means of approved flyers posted in selected PHCs. Interested WLA will approach the research staff, stationed at the PHC to be screened for eligibility via a consent script. Once eligibility is determined for the WLA, based upon the following criteria: age, HIV and ART status (validated by ART and HIV card); having a child (3-8 years) and whether or not the WLA was a participant of the previous intervention group from the Asha pilot study, a parental consent will be obtained from the WLA for permission to include her oldest child in the study. The oldest child between 3-8 years of age will be brought in to the research office or PHC (after mother speaks with the child at home). All children will have blood work drawn and physical health assessment on their first visit (total of 15 minutes). All eligible WLA will undergo a second consent for enrollment. General Procedure: Following informed consent, the WLA will be randomly assigned into one of four programs 1) Asha Support Only; 2) Asha Support + Training; 3) Asha Support + Food; or 4) Asha Support + Training + Food. After blood draw and physical assessment of the WLA, an appointment will be made for the assigned interviewer (blinded to program) to visit the WLA at their home preferably (or other location of choice) to conduct several 24 hour dietary assessments. Urine will be collected in labeled bottles on the morning after the 3rd day of the diet recall by the interviewer and sent directly to the lab in a cooler. Also, on the same day, the baseline assessment will be entered into the PC tablets; 50 minutes estimated with breaks). After a longer break, the WLA will then be asked to respond to additional questions about the sociodemographic and psychomotor development of their child (about 30 minutes). Interviewers will visit the WLA monthly until the end of the intervention (month 6) to provide individual weekly Asha Support and conduct group sessions and collect ongoing data, 24-hour recall, and ART pill count for WLA, and follow up questionnaires at 6-, 12- and 18-months.

DETAILED DESCRIPTION:
Rural women living with AIDS (WLA) in India continue to face profound challenges in accessing and following treatment regimens, caring for family members, and maintaining positive mental health. Furthermore, they are generally underweight and malnourished, with adherence to antiretroviral therapy (ART) at levels lower than 50%. While the Indian Government's National Rural Health Mission utilizes a successful model to address the health needs of the rural population by training village women as Ashas (Accredited Social Work Activists) to enhance health of pregnant women and their infants, the focus on rural WLA needs to be significantly strengthened. U.S. and Indian collaborators recently completed an R34 pilot study which has demonstrated successful improvement in ART adherence, CD4 levels, and physical and mental health among rural Indian WLA. In total, 34 rural intervention WLA were supported by grant-trained, HIV-focused Ashas who provided assistance to WLA in decreasing barriers to ART adherence and provided protein supplementation compared to equal numbers of usual care WLA who received minimal protein supplementation. While very successful, our Asha pilot study monitored only WLA, despite the fact that many rural children are also at risk for delayed physical growth and psychomotor development. More importantly, we were not able to separate the nutritional component from the care and support component of the Asha, did not incorporate nutritional biomarkers, and were limited by only a six-month follow-up. In light of the mandate to advance both the science of nutrition and sustainability in real settings, our experienced team proposes to build on and extend our successful pilot work to meet this need, by assessing the incremental advantages of nutritional support to Asha care and support alone, and the impact of these programs on an index child (oldest between 3-8 years). In addition, we will take advantage of rural India's excellent mobile phone coverage and computer technology for both wireless data collection and data transfer. The proposed longitudinal study will use a 2x2 factorial design, specifically, 1) Asha support alone for WLA , vs. 2) Asha support for WLA + nutrition (food-based) training, vs. 3) Asha support for WLA + food supplementation, vs. 4) Asha support for WLA + nutrition training + food supplementation, to test the effects of nutrition training and/or food supplementation on primary outcomes of anthropometric parameters and immune status (CD4 levels) of the WLA at 6-, 12- and 18-month follow-up; and secondarily on ART adherence, psychological health, nutritional adequacy and lipid status of the WLA over time. Based upon reviewers' comments, among index children, we streamlined our assessments to include anthropometric parameters and psychomotor development; and among those HIV positive, immune status.

ELIGIBILITY:
Inclusion Criteria: 1) WLA, 18-50 years of age; 2) receiving Antiretroviral Therapy (ART) for > three months; validated by an ART card given by the district hospital to all ART patients; 3) Blood Cell count > 100 validated by HIV card given by district hospital; 4) reporting to have a child aged 3-8 living with them; 5) not involved in Asha Life Intervention group of the first Asha study -

Exclusion Criteria: WLA not between the ages of 18 to 50; not on Antiretroviral Therapy (ART) for at least three months and has a blood cell count of less than 100; reporting no children between the ages of 3 to 8; and a previous participant of the Asha Life Intervention group of the first Asha study.

-

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 600 (Actual)
Dates: Start 2013-08; Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Change in weight | 6-, 12- and 18-month followup
  Weight gain as measured in BMI (kg/m2)
Change in CD4+ T cell count | 6-, 12- and 18-month followup
  Measure of immune status in cells/mm3
Change in muscle mass | 6-, 12- and 18-month followup
  Measured by the Bioelectrical Impedance (BIA)

SECONDARY OUTCOMES:
Change in ART adherence | 6-, 12- and 18-month followup
  Measured by visual analog scale
Change in depressive symptomatology | 6-, 12- and 18-month followup
  Measured by Center for Epidemiologic Studies Depression Scale (CES-D)
Change in internalized stigma | 6-, 12- and 18-month followup
  Measured by the Internalized Stigma Scale
Change in nutritional adequacy | 6-, 12- and 18-month followup
  Nutritional adequacy of the WLA over 18 months, measured by comparisons of vitamin, mineral and macronutrient intake, guided by dietary recommendations
Change in lipid normalization | 6-, 12- and 18-month followup
  Lipid normalization of WLA (triglycerides and cholesterol)
Change in anthropometric parameters and psychomotor development of the index children | 6-, 12- and 18-month followup
  Anthropometric parameters and psychomotor development of the index children at 6-12-, and 18-month follow-up; among those HIV-infected, we will also assess CD4 levels over time.

CONTACTS AND LOCATIONS:
Overall Officials: Adeline M Nyamathi, PhD, Principal Investigator — UCI Sue & Bill Gross School of Nursing; Maria Ekstrand, PhD, Principal Investigator — University of California, San Francisco; Sanjeev Sinha, MD, Principal Investigator — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences (AIIMS), New Delhi, India

REFERENCES:
- [Background] Nyamathi A, Ekstrand M, Srivastava N, Carpenter CL, Salem BE, Al-Harrasi S, Ramakrishnan P, Sinha S. ASHA-Life Intervention Perspectives Voiced by Rural Indian Women Living With AIDS. Health Care Women Int. 2016;37(4):412-25. doi: 10.1080/07399332.2015.1066790. Epub 2015 Jul 6. PMID 26147930
- [Background] Srivastava N, Nyamathi AM, Sinha S, Carpenter C, Satyanarayana V, Ramakrishna P, Ekstrand M. Women living with AIDS in rural Southern India: Perspectives on mental health and lay health care worker support. J HIV AIDS Soc Serv. 2017;16(2):170-194. doi: 10.1080/15381501.2016.1274703. Epub 2017 Feb 23. PMID 29056879
- [Background] Salem BE, Bustos Y, Shalita C, Kwon J, Ramakrishnan P, Yadav K, Ekstrand ML, Sinha S, Nyamathi AM. Chronic Disease Self-Management Challenges among Rural Women Living with HIV/AIDS in Prakasam, Andhra Pradesh, India: A Qualitative Study. J Int Assoc Provid AIDS Care. 2018 Jan-Dec;17:2325958218773768. doi: 10.1177/2325958218773768. PMID 29756550
- [Result] Nyamathi A, Ekstrand M, Heylen E, Ramakrishna P, Yadav K, Sinha S, Hudson A, Carpenter CL, Arab L. Relationships Among Adherence and Physical and Mental Health Among Women Living with HIV in Rural India. AIDS Behav. 2018 Mar;22(3):867-876. doi: 10.1007/s10461-016-1631-3. PMID 27990577
- [Result] Nyamathi AM, Ekstrand M, Yadav K, Ramakrishna P, Heylen E, Carpenter C, Wall S, Oleskowicz T, Arab L, Sinha S. Quality of Life Among Women Living With HIV in Rural India. J Assoc Nurses AIDS Care. 2017 Jul-Aug;28(4):575-586. doi: 10.1016/j.jana.2017.03.004. Epub 2017 Mar 24. PMID 28473182
- [Result] Shin SS, Carpenter CL, Ekstrand ML, Yadav K, Shah SV, Ramakrishnan P, Pamujula S, Sinha S, Nyamathi AM. Household Food Insecurity as Mediator of the Association Between Internalized Stigma and Opportunistic Infections. AIDS Behav. 2018 Dec;22(12):3897-3904. doi: 10.1007/s10461-018-2193-3. PMID 29934793
- [Result] Ekstrand ML, Heylen E, Mazur A, Steward WT, Carpenter C, Yadav K, Sinha S, Nyamathi A. The Role of HIV Stigma in ART Adherence and Quality of Life Among Rural Women Living with HIV in India. AIDS Behav. 2018 Dec;22(12):3859-3868. doi: 10.1007/s10461-018-2157-7. PMID 29789984
- [Derived] Nyamathi AM, Carpenter CL, Ekstrand ML, Yadav K, Garfin DR, Muniz LC, Kelley M, Sinha S. Randomized controlled trial of a community-based intervention on HIV and nutritional outcomes at 6 months among women living with HIV/AIDS in rural India. AIDS. 2018 Nov 28;32(18):2727-2737. doi: 10.1097/QAD.0000000000002016. PMID 30289802